CLINICAL TRIAL: NCT04149275
Title: A Phase II Single Arm Study of Cabozantinib Plus Nivolumab and Ipilimumab in Women With Recurrent Gynecologic Carcinosarcoma
Brief Title: Cabozantinib Plus Nivolumab and Ipilimumab in Women With Recurrent Gynecologic Carcinosarcoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding withdrawn by sponsor
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Rebecca Arend, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300003948
Record Dates: First submitted 2019-10-22; First posted 2019-11-04 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Carcinosarcoma of Ovary; Carcinosarcoma of Uterus; Carcinosarcoma of Vagina
Keywords: Cabozantinib; Nivolumab; Ipilimumab; tyrosine-kinase inhibitor; anti-PD-1; anti-CTLA-4
MeSH Terms: interventions — cabozantinib; Tyrosine Kinase Inhibitors; Ipilimumab; Nivolumab; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cabozantinib + Nivolumab + Ipilimumab (Experimental): All recurrent carcinosarcomas
  Interventions: Drug: Cabozantinib; Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Cabozantinib — Treatment with oral Cabozantinib once daily
  Other Names: tyrosine kinase inhibitor
Drug: Ipilimumab — IV administration of Ipilimumab on 21 day cycles
  Other Names: anti-CTLA-4
Drug: Nivolumab — IV administration of Nivolumab on 21 day cycles, followed by Nivolumab maintenance on 28 day cycles
  Other Names: anti-PD-1

SUMMARY:
The purpose of this study is to test the safety of Cabozantinib in combination with Nivolumab and Ipilimumab and see what affects that this combination treatment has on those with recurrent carcinosarcomas.

DETAILED DESCRIPTION:
Primary Objectives:

• To estimate the proportion of patients with recurrent carcinosarcoma, who survive progression-free for at least 6 months, treated with cabozantinib + nivolumab + ipilimumab in the second-line and beyond setting (per iRECIST).

Secondary Objectives:

* To evaluate time to progression (Time Frame: From the date the patient received the first study treatment dose until the date of first documented progression, assessed up to 2 years). Progression Free Survival (PFS) according to iRECIST.
* To determine the nature and degree of toxicity of cabozantinib + nivolumab + ipilimumab in this cohort of patients. Toxicity according to CTCAE v4.03
* To estimate the overall survival (OS) of patients with carcinosarcoma treated with cabozantinib + nivolumab + ipilimumab

Exploratory Objectives:

* To determine expression of biomarkers, which will include PD-L1 and MET expression by IHC, MSI status by NGS, and other relevant potential biomarkers.
* To determine whether these marker expression levels alone or in combination are associated with response, PFS, and/or overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of carcinosarcoma (independent of organ of origin).
2. Received at least one prior chemotherapy regimen for their cancer.
3. Must have measurable or evaluable lesion defined by iRECIST.
4. Recovery to baseline or ≤ Grade 1 CTCAE v4 from toxicities related to any prior treatments, unless AE(s) are clinically non-significant and/or stable on supportive therapy.
5. Karnofsky performance status greater than or equal to 70% or ECOG PS = 0~2
6. Age ≥ 18 years.
7. Adequate organ and marrow function, based upon meeting all of the following laboratory criteria within 14 days before first dose of study treatment:

   1. Absolute neutrophil count (ANC) ≥ 1500/mm3 (≥ 1.5 GI/L) without granulocyte colony-stimulating factor support.
   2. White blood cell count ≥ 2500/mm3 (≥ 2.5 GI/L).
   3. Platelets ≥ 100,000/mm3 (≥ 100 GI/L) without transfusion.
   4. Hemoglobin ≥ 9 g/dL (≥ 90 g/L).
   5. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) ≤ 3 x upper limit of normal (ULN). ALP ≤ 5 x ULN with documented bone metastases.
   6. Total bilirubin ≤ 1.5 x ULN (for subjects with Gilbert's disease ≤ 3 x ULN).
   7. Serum albumin ≥ 2.8 g/dl.
   8. Serum creatinine ≤ 2.0 x ULN or calculated creatinine clearance ≥ 30 mL/min (≥ 0.5 mL/sec) using the Cockcroft-Gault equation: [(140 - age) x weight (kg)/(serum creatinine [mg/dL] × 72)] × 0.85
   9. Urine protein/creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.2 mg/mmol).
8. Capable of understanding and complying with the protocol requirements and must have signed the informed consent document.
9. Women of childbearing potential (WOCBP) ie. sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (eg, barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 5 months after the last dose of study treatment.
10. Females should not breastfeed while receiving treatment on trial.
11. Female subjects of childbearing potential must not be pregnant at screening. Females of childbearing potential are defined as premenopausal females capable of becoming pregnant (ie, females who have had any evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy). However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, low body weight, ovarian suppression or other reasons.

Exclusion Criteria:

1. Prior treatment with cabozantinib.
2. Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks before first dose of study treatment.
3. Receipt of any type of cytotoxic, biologic or other systemic anticancer therapy (including investigational) within 4 weeks before first dose of study treatment.
4. Radiation therapy for bone metastasis within 2 weeks, any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before the first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.
5. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before first dose of study treatment. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of first dose of study treatment.
6. Concomitant anticoagulation with oral anticoagulants (eg, warfarin, direct thrombin and Factor Xa inhibitors) or platelet inhibitors (eg, clopidogrel). Allowed anticoagulants are the following:

   1. Low-dose aspirin for cardioprotection (per local applicable guidelines) is permitted.
   2. Low-dose low molecular weight heparins (LMWH) are permitted.
   3. Anticoagulation with therapeutic doses of LMWH is allowed in subjects without known brain metastases who are on a stable dose of LMWH for at least 6 weeks before first dose of study treatment, and who have had no clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.
7. The subject has prothrombin time (PT)/INR or partial thromboplastin time (PTT) test ≥ 1.3 x the laboratory ULN within 7 days before the first dose of study treatment.
8. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

   a. Cardiovascular disorders: i. Congestive heart failure New York Heart Association Class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias.

   ii. Uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mm Hg systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment.

   iii. Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (eg, deep venous thrombosis, pulmonary embolism) within 6 months before first dose.

   b. Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation: i. The subject has evidence of tumor invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (eg, Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction.

   ii. Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose.

   Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose.

   c. Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (eg, pulmonary hemorrhage) within 12 weeks before first dose.

   d. Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation.

   e. Lesions invading or encasing any major blood vessels. f. Other clinically significant disorders that would preclude safe study participation.

   i. Serious non-healing wound/ulcer/bone fracture. ii. Uncompensated/symptomatic hypothyroidism. iii. Moderate to severe hepatic impairment (Child-Pugh B or C).
9. Major surgery (eg, GI surgery, removal or biopsy of brain metastasis) within 8 weeks before first dose of study treatment. Complete wound healing from major surgery must have occurred 1 month before first dose and from minor surgery (eg, simple excision, tooth extraction) at least 10 days before first dose. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
10. Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms per electrocardiogram (ECG) within 28 days before first dose of study treatment [add reference for Fridericia formula].

    Note: If a single ECG shows a QTcF with an absolute value > 500 ms, two additional ECGs at intervals of approximately 3 min must be performed within 30 min after the initial ECG, and the average of these three consecutive results for QTcF will be used to determine eligibility.
11. Inability to swallow tablets.
12. Previously identified allergy or hypersensitivity to components of the study treatment formulations.
13. Diagnosis of another malignancy within 2 years before first dose of study treatment, except for superficial skin cancers, or localized, low grade tumors deemed cured and not treated with systemic therapy.
14. Patients with concurrent cytotoxic chemotherapy or radiation therapy are excluded.
15. Patients with a serious chronic or acute illness, such as cardiac disease (NYHA class III or IV), hepatic disease, or other illness considered by the Principal Investigator as unwarranted high risk for investigational drug treatment.
16. Patients with a medical or psychological impediment to probable compliance with the protocol should be excluded.
17. Presence of a known active acute or chronic infection including: a urinary tract infection, HIV or viral hepatitis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Percent progression free survival according to RECIST v1.1 | Baseline through 6 months
  To estimate the proportion of patients with recurrent carcinosarcoma, who survive progression-free for at least 6 months, treated with cabozantinib + nivolumab + ipilimumab in the second-line and beyond setting (per iRECIST).

SECONDARY OUTCOMES:
Percent time to progression according to RECIST v1.1 | Baseline through 2 years
  To evaluate time to progression (Time Frame: From the date the patient received the first study treatment dose until the date of first documented progression, assessed up to 2 years). Progression Free Survival (PFS) according to iRECIST.
Percent overall survival according to RECIST v1.1 | Baseline through 2 years
  To estimate the overall survival (OS) of patients with carcinosarcoma treated with cabozantinib + nivolumab + ipilimumab
Percent of patients with toxicity according to CTCAE v4.03 | Baseline through 2 years
  To determine the nature and degree of toxicity of cabozantinib + nivolumab + ipilimumab in this cohort of patients. Toxicity according to CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca C Arend, MD, MSPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
To Be Determined